CLINICAL TRIAL: NCT06804824
Title: A Phase 1/1b, Open-Label, Multicenter, First-in-Human Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Anti-Tumor Activity of VVD-159642, a RAS-PI3Kα Inhibitor, as a Single Agent and in Combination in Participants With Advanced Solid Tumors
Brief Title: A First-in-Human (FIH) Study to Evaluate the Safety and Tolerability of VVD-159642 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vividion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VVD-159642-01
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: RAS; PI3K; KRAS; MEK; Phase I; solid tumors; KRAS G12C; HER2
MeSH Terms: interventions — sotorasib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Dose Escalation: VVD-159642 Single Agent (Experimental): Participants will receive ascending doses of VVD-159642, orally, daily in 21-day treatment cycles during Part 1.
  Interventions: Drug: VVD-159642
- Part 2: Dose Expansion (Cohort A): VVD-159642 Single Agent (Experimental): Participants will receive VVD-159642 at the recommended dose for expansion (RDE), orally, daily in 21-day treatment cycles during Part 2.
  Interventions: Drug: VVD-159642
- Part 2: Dose Expansion (Cohort B): VVD-159642 + Sotorasib (Experimental): Participants will receive VVD-159642 at RDE orally, daily in combination with sotorasib, in 21-day treatment cycles after a safety run-in.
  Interventions: Drug: VVD-159642; Drug: Sotorasib
- Part 2: Dose Expansion (Cohort C): VVD-159642 + Trametinib (Experimental): Participants will receive VVD-159642 at RDE orally, daily in combination with trametinib, in 21-day treatment cycles after a safety run-in.
  Interventions: Drug: VVD-159642; Drug: Trametinib

INTERVENTIONS:
Drug: VVD-159642 — Oral capsules
Drug: Sotorasib — Oral tablets
  Arms: Part 2: Dose Expansion (Cohort B): VVD-159642 + Sotorasib
Drug: Trametinib — Oral tablets
  Arms: Part 2: Dose Expansion (Cohort C): VVD-159642 + Trametinib

SUMMARY:
A FIH study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary anti-tumor activity of VVD-159642, a rat sarcoma viral oncogene-phosphatidylinositol 3-kinase alpha (RAS-PI3Kα) inhibitor, as a single agent and in combination with either sotorasib or trametinib in participants with advanced solid tumors.

ELIGIBILITY:
Key Inclusion Criteria:

* For Part 1 Dose Escalation, the prospective participant must have histologically confirmed pancreatic ductal adenocarcinoma (PDAC), colorectal cancer (CRC), non-small cell lung cancer (NSCLC), or any solid tumor that harbors a rat sarcoma viral oncogene (RAS) alteration [Kirsten rat sarcoma viral oncogene homolog (KRAS), neuroblastoma RAS viral oncogene homolog (NRAS), Harvey rat sarcoma viral oncogene homolog (HRAS)] as per local /historical testing; any solid tumor that harbors an epidermal growth factor receptor (EGFR) alteration as per local/historical testing; or human epidermal growth factor receptor 2 (HER2) overexpression (immunohistochemistry [IHC] 3+ or IHC 2+/fluorescence in situ hybridization [FISH] positive) as per local/historical testing.
* Have histologically or cytologically confirmed metastatic or unresectable solid tumors.
* Measurable disease by RECIST version 1.1 as assessed by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Adequate bone marrow, kidney, and liver function as defined in the protocol.
* Able to take oral medications.

Key Exclusion Criteria:

* Active central nervous system (CNS) malignancies.
* History of cardiac diseases as defined in detail in the protocol.
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's opinion).
* History of inflammatory bowel disease or any malabsorption syndrome or any conditions that would interfere with enteral absorption and/or may interfere with the conduct of the study.
* Active hepatitis B infection [positive for hepatitis B surface antigen and Hepatitis B virus deoxyribonucleic acid (DNA)].
* Active hepatitis C infection (positive anti-hepatitis C virus [HCV] antibody and quantitative HCV ribonucleic acid (RNA) results greater than the lower limits of detection of the assay).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence and Severity of Dose-limiting Toxicities (DLTs) | From Day 1 to Day 21 of Cycle 1 [cycle length=21 days]
Part 2: Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 29 months
Part 2: Incidence and Severity of Clinically Significant Changes in Vital Signs | Up to approximately 29 months
Part 2: Incidence and Severity of Clinically Significant Changes in Laboratory Evaluations | Up to approximately 29 months

SECONDARY OUTCOMES:
Part 1: Recommended Dose for Expansion (RDE) of VVD-159642 as a Single Agent | Up to approximately 29 months
  The RDE will be based on safety, tolerability, PK, and preliminary anti-tumor activity of VVD-159642 as a single agent during the dose escalation phase.
Part 2: Recommended Phase 2 Dose (RP2D) of VVD-159642 as a Single Agent and in Combination with Sotorasib and Trametinib | Up to approximately 29 months
  The RP2D will be based on safety, tolerability, PK and preliminary anti-tumor activity of VVD-159642 as single agent, and in combination with sotorasib and trametinib during Part 2.
Part 2: Overall Response Rate (ORR) | Up to approximately 29 months
  ORR is defined as the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator assessment.
Part 2: Duration of Response (DoR) | Up to approximately 29 months
  DOR is defined as the time from initial response of CR or PR to progressive disease or death, whichever comes first per RECIST version 1.1 by investigator assessment.
Part 2: Progression-free Survival (PFS) | Up to approximately 29 months
  PFS is defined as the time from the date of randomization to the time of confirmed disease progression or death, whichever occurs first per RECIST version 1.1 by investigator assessment.
Part 2: Disease Control Rate (DCR) | Up to approximately 29 months
  DCR is defined as the percentage of participants achieving CR or PR, or stable disease (SD) per RECIST version 1.1 by investigator assessment.
Parts 1 and 2: Area Under the Plasma Concentration-time Curve (AUC) of VVD-159642 as a Single Agent and in Combination With Sotorasib and Trametinib | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)
Parts 1 and 2: Maximum Plasma Concentration (Cmax) of VVD-159642 as a Single Agent and in Combination With Sotorasib and Trametinib | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)
Parts 1 and 2: Half-life (t1/2) of VVD-159642 as a Single Agent and in Combination With Sotorasib and Trametinib | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - START Mid West, Grand Rapids, Michigan
  - NEXT Austin, Austin, Texas
  - NEXT Dallas, Irving, Texas
  - START San Antonio, San Antonio, Texas
  - NEXT San Antonio, San Antonio, Texas
  - START Mountain, Ogden, Utah
  - NEXT Virginia, Fairfax, Virginia
- Australia (2):
  - Clinical Research South Australia (CRSA), Adelaide, South Australia
  - Linear Clinical, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No